CLINICAL TRIAL: NCT01569867
Title: An Observational Study Investigating Genetic Influences on Statin Plasma Concentrations in Adult African American Patients
Brief Title: Genetic Influences on Statin Blood Concentrations in African Americans
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Sakima Smith, Associate Professor, Ohio State University
Other Study IDs: OSU 2011H0402; K23GM100372 (NIH); R01MD011307 (NIH)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Hyperlipidemia; Hypercholesterolemia; Dyslipidemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen plasma and frozen nuclear pellet
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- statin

SUMMARY:
This study intends to determine the effects of genetic polymorphisms on statin response and daily systemic exposure (24-hour area under the time-concentration curve) of statins in African-American patients.

ELIGIBILITY:
Inclusion Criteria:

* African-American patients taking a statin metabolized by CYP3A (e.g., atorvastatin, simvastatin, or lovastatin)

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals will be recruited from various hospitals, ancillary clinics, and primary-care offices affiliated with the Ohio State University Medical Center (OSUMC).
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
24-hour area under the time-concentration curve of statin concentrations in plasma | 2 years

SECONDARY OUTCOMES:
Incidence of statin-associated muscle symptoms (SAMS) | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Kitzmiller, MD PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Wang J, Luzum JA, Phelps MA, Kitzmiller JP. Liquid chromatography-tandem mass spectrometry assay for the simultaneous quantification of simvastatin, lovastatin, atorvastatin, and their major metabolites in human plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2015 Mar 1;983-984:18-25. doi: 10.1016/j.jchromb.2014.12.029. Epub 2015 Jan 13. PMID 25612772